CLINICAL TRIAL: NCT05775159
Title: A Phase II, Open-Label, Multi-Drug, Multi-Center, Master Protocol to Evaluate the Efficacy and Safety of Novel Immunomodulators as Monotherapy and in Combination With Anticancer Agents in Participants With Advanced Hepatobiliary Cancer (GEMINI-Hepatobiliary)
Brief Title: Study of Novel Immunomodulators as Monotherapy and in Combination With Anticancer Agents in Participants With Advanced Hepatobiliary Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7987C00001
Record Dates: First submitted 2023-03-02; First posted 2023-03-20 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer
Keywords: Hepatobiliary cancer; Hepatocellular carcinoma; Biliary tract cancer; GEMINI-Hepatobiliary; MEDI5752; AZD2936; Bispecific antibody; Volrustomig; Rilvegostomig
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms | interventions — Bevacizumab; lenvatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1A (Experimental): Volrustomig monotherapy
  Interventions: Drug: Volrustomig
- Cohort 1B (Experimental): Volrustomig combination with bevacizumab
  Interventions: Drug: Volrustomig; Drug: Bevacizumab
- Cohort 1C (Experimental): Volrustomig combination with lenvatinib
  Interventions: Drug: Volrustomig; Drug: Lenvatinib
- Cohort 2A (Experimental): Rilvegostomig combination with Gemcitabine and Cisplatin
  Interventions: Drug: Rilvegostomig; Drug: Gemcitabine; Drug: Cisplatin
- Cohort 2B (Experimental): Volrustomig combination with Gemcitabine and Cisplatin
  Interventions: Drug: Volrustomig; Drug: Gemcitabine; Drug: Cisplatin
- Cohort 1D (Experimental): Volrustomig combination with rilvegostomig and bevacizumab
  Interventions: Drug: Volrustomig; Drug: Bevacizumab; Drug: Rilvegostomig
- Cohort 1E (Experimental): Rilvegostomig combination with bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Rilvegostomig

INTERVENTIONS:
Drug: Volrustomig — CTLA-4/Anti-PD-1 Bispecific Antibody
  Arms: Cohort 1A; Cohort 1B; Cohort 1C; Cohort 1D; Cohort 2B
Drug: Bevacizumab — 15 mg/kg, IV (in the vein) on day 1 of each 21 day cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Arms: Cohort 1B; Cohort 1D; Cohort 1E
Drug: Lenvatinib — Daily use per oral (8 mg capsules/day for participants < 60 kg or 12 mg/day for participants ≥ 60 kg) of 21 day cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Arms: Cohort 1C
Drug: Rilvegostomig — anti- PD-1 and TIGIT bispecific antibody
  Arms: Cohort 1D; Cohort 1E; Cohort 2A
Drug: Gemcitabine — 1000 mg/m2, IV infusion
  Arms: Cohort 2A; Cohort 2B
Drug: Cisplatin — 25 mg/m2, IV infusion
  Arms: Cohort 2A; Cohort 2B

SUMMARY:
GEMINI-Hepatobiliary study will assess the efficacy, safety and tolerability of novel immunomodulators alone and in combination with other anticancer drugs in participants with specified advanced solid tumors.

DETAILED DESCRIPTION:
This Phase II, open-label, uncontrolled, multicentre study evaluating the preliminary efficacy and safety of Volrustomig or Rilvegostomig as monotherapy (MONO) and/or in combination with anticancer agents (COMBO) in participants with advanced hepatobiliary cancer (e.g., HCC, BTC, etc.).

This study has a modular design with independent substudies. In Substudy 1, Volrustomig and Rilvegostomig will be evaluated as monotherapy and/or in combination with other anticancer drugs in approximately 200 evaluable participants with advanced HCC.

In Substudy 2, the efficacy and safety of Rilvegostomig or Volrustomig plus gemcitabine and cisplatin are investigated in approximately 90 evaluable participants with advanced BTC who have not received previous treatment for advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the ICF.
* Provision of a signed and dated written ICF.
* Confirmed locally advanced or metastatic solid tumor specified in substudy based on histopathology.
* Adequate organ and bone marrow function.
* At least 1 measurable not previously irradiated lesion per RECIST 1.1
* Life expectancy of at least 12 weeks at the time of screening.
* Willing and able to provide an adequate tumor sample.

Exclusion Criteria:

* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders.
* Uncontrolled intercurrent illness.
* History of another primary malignancy, leptomeningeal carcinomatosis, and active primary immunodeficiency.
* Active infection, brain metastases or spinal cord compression.
* Participants co-infected with HBV and hepatitis D virus (HDV).
* Previous treatment in the present study.
* For substudy 1, history of hepatic encephalopathy within 12 months prior to treatment allocation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 years
  ORR is defined as the proportion of participants who have a confirmed CR (complete response) or confirmed PR (partial response), determined by the Investigator at local site per RECIST 1.1 (For HCC sub-study 1)
The number of participants with adverse events/serious adverse events | Through study completion, an average of 2 years
  Number of participants with adverse events and with serious adverse events including abnormal clinical observations, abnormal Electrocardiogram (ECG) parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline.
Progression free survival (PFS) | Through study completion, an average of 2 years
  PFS is defined as the time from the start of studyintervention until progression per RECIST 1.1 as assessed by the Investigator at the local site or death due to any cause in the absence of progression, whichever occurs first. (For BTC sub-study 2)

SECONDARY OUTCOMES:
Duration Of Response (DOR) | Through study completion, an average of 2 years
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 by the Investigator at local site or death due to any cause in the absence of disease progression, whichever occurs first.
Disease Control Rate (DCR) | At 12 and 24 weeks
  DCR at 12 and 24 weeks is defined as the percentage of participants who have a Complete response (CR) or Partial response (PR) in the first 13 and 25 weeks or who have Stable disease (SD) for at least 11 and 23 weeks after the date of first dose respectively, per RECIST 1.1 as assessed by the investigator at local site and derived from the raw tumour data.
Progression free survival (PFS) | Through study completion, an average of 2 years
  PFS is defined as the time from the start of study intervention until progression per RECIST 1.1 as assessed by the Investigator at the local site or death due to any cause in the absence of progression, whichever occurs first.
Overall Survival (OS) | Through study completion, an average of 2 years
  OS is defined as the time from the start of study intervention until the date of death due to any cause, whichever occurs first.
Anti Drug Antibody (ADA) | Through study completion, an average of 2 years
  Incidences of ADAs against novel immunomodulators in serum.
Pharmacokinetics of novel immunomodulators: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the administration of novel immunomodulators ( approx 2 years )
  Maximum observed plasma concentration of the study drug
Pharmacokinetics of novel immunomodulators: Time to maximum plasma concentration of the study drug (T-max) | From the first dose of study intervention, at predefined intervals throughout the administration of novel immunomodulators ( approx 2 years )
  Time to maximum observed plasma concentration of the study drug
lmmunogenicity of novel immunomodulators | From the first dose of study intervention, at predefined intervals throughout the administration of novel immunomodulators ( approx 2 years)
  The number and percentage of participants who develop ADAs.
Objective response rate (ORR) | Through study completion, an average of 2 years
  ORR is defined as the proportion of participants who have a confirmed CR (complete response) or confirmed PR (partial response), determined by the Investigator at local site per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (47):
- United States (10):
  - Research Site, Birmingham, Alabama
  - Research Site, Costa Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Miami Beach, Florida
  - Research Site, Dyer, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, New York, New York
  - Research Site, Dallas, Texas
  - Research Site, Fairfax, Virginia
- China (13):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Italy (4):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rozzano
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Yokohama
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Liuying
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home